CLINICAL TRIAL: NCT04218344
Title: The Harefield Acute Myocardial Infarction Cohort
Acronym: HEART - ACS
Status: Recruiting | Type: Observational
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS ID - 25908
Record Dates: First submitted 2020-01-02; First posted 2020-01-06 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood, 60mls per participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute Coronary Syndrome - Iscaemia: Patients who present with chest pain, undergo emergency angiogram and receive a cardiac stent.
  Interventions: Other: 60mls of blood donated for research analysis
- Acute Coronary Syndrome - Non-Ischaemic: Patients who present with chest pain but angiography reveals normal coronary arteries.
  Interventions: Other: 60mls of blood donated for research analysis

INTERVENTIONS:
Other: 60mls of blood donated for research analysis — All patients presenting with a possible Acute Coronary Syndrome will be invited to donate 60 mls of blood at the time of their angiogram.

SUMMARY:
In this project the investigator's plan to collect blood during a patient's routine angiogram procedure which they will have due to having suffered a heart attack. Data from the patients' routine procedures for this condition, including but not exclusively, ECG, Echocardiogram, MRI scans, will be collected. The aim of the research project is to analyse the blood samples and identify novel biomarkers and clinical parameters associated with acute coronary syndromes. The investigator's will particularly focus on markers of inflammation and micro-organism activity. The investigator's hope that this will help to gain more knowledge about what causes heart disease and how various conditions can be treated more efficiently. The investigator's will follow-up and collect further research data via a questionnaire at the routine 6 weeks and 6 months follow-up appointment after the angiogram procedure. Participants will also be telephoned at one-year post procedure, to update any events and medication status and data will thereafter be collected form data held by the hospital without having to contact the participant. Remaining blood samples will be stored securely for further analysis into blood and other markers.

DETAILED DESCRIPTION:
Acute coronary syndromes (ACS), i.e. patients presenting with ST-segment elevation myocardial infarction (STEMI), non ST-segment elevation myocardial infarction (non-STEMI) or unstable angina, are still a major cause of morbidity and mortality in the United Kingdom and beyond. In spite of the enormous progress made in the last decades, the in hospital mortality has plateaued recently, and the event rate after the infarction is still high with one in 8 patients having a second event (i.e. death, myocardial infarction, heart failure, revascularization among others) within a year of follow-up.

After the acute event, risk stratification is important and will be come even more sophisticated than it currently is with the advent of anatomic risk scores (SYNTAX II Score), novel biomarkers and novel drugs allowing for more precise characterization of the patients individual risk and more tailored secondary prevention strategies (Precision Medicine).

Indeed, particularly the upcoming treatment strategies with bio-logicals (i.e. monoclonal antibodies, e.g. against PCSK9) and genetic tools (i.e. RNA interference, antisense technology) will require precise risk assessment for cost-effective use of these promising new tools.

It is anticipated that this study will help the investigator's to describe the heart attack population in a robust manner with a wealth of clinical data as well as blood samples for bio-markers.

ELIGIBILITY:
Inclusion Criteria:

• All patients presenting to Harefield Hospital through the Primary Percutaneous Coronary Intervention programme, with ST-segment elevation myocardial infarction, non ST-segment elevation myocardial infarction, unstable angina, Tako Tsubo syndrome, spontaneous coronary artery dissection and acute myocarditis, with the intention to assess with coronary angiography.

Exclusion Criteria:

* Patients will be able to self-exclude if they do not provide full informed consent
* Every effort will be made to obtain informed consent from all patients.
* Patients who do not survive the hospital episode will undergo a Professional or Personal Consultee process of assumed consent.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients presenting to Harefield Hospital through the Primary Percutaneous Coronary Intervention programme
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-01-09 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
To identify novel biomarkers and clinical parameters associated with acute coronary syndromes caused by coronary artery disease | 2 - 5 Years
  1. Inflammatory markers
  2. Microbiome metabolites

SECONDARY OUTCOMES:
To define the patient population with Myocardial Infarction with Non-Obstructive Coronary Artery disease (MINOCA) and determine the individual risks of these patients (eg. TakoTsubo Syndrome and Acute Myocarditis). | 2 - 5 Years
  To define the patient population with Myocardial Infarction with Non-Obstructive Coronary Artery disease (MINOCA) and determine the individual risks of these patients (eg. TakoTsubo Syndrome and Acute Myocarditis).
To explore the concept of personalised medicine for future patients, based on the identification of novel biomarkers. | 2 - 5 Years
  To explore the concept of personalised medicine for future patients, based on the identification of novel biomarkers.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Harefield Hospital, Harefield, Middlesex
  - Royal Brompton and Harefield NHS Foundation Trust, Uxbridge, Middlesex

IPD SHARING:
Plan to Share IPD: No